CLINICAL TRIAL: NCT07119762
Title: Effects of a 20-week Combined Mat-Pilates Training With Dual Task Exercise for Improving Trunk Strength and Stability, Balance, Cognitive Function, and Risk of Falls in Older Adults.
Brief Title: Effects of 20-week Mat-Pilates & Dual-Task Training on Strength, Balance, Cognition, and Fall Risk in Older Adults
Acronym: Pilates&ST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CEFADE 41_2022; 2023.02364.BD (Other Grant/Funding Number: FCT: Fundação para a Ciências e Tecnlogia)
Record Dates: First submitted 2025-08-05; First posted 2025-08-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-05

CONDITIONS: Healthy People Programs
Keywords: AGING.; PHYSICAL EXERCISE; CORE STRENGTH; STABILITY
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Physical activity intervention (Pilates)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates (Experimental): depois
  Interventions: Other: Pilates sections
- Control Group (No Intervention)

INTERVENTIONS:
Other: Pilates sections — This intervention combines Pilates with dual-task training over 20 weeks, featuring twice-weekly 60-minute sessions at moderate to vigorous intensity. It is uniquely grounded in methods from the Polestar and PhysicalMind schools and adapted for older adults (≥65 years), utilizing chairs, elastic bands, and minimal equipment. Unlike typical exercise programs, this protocol integrates cognitive tasks within Pilates exercises to simultaneously challenge physical and executive functions. Exercise intensity is individualized using heart rate monitors and the Borg scale. Assessments include trunk strength (Biodex System 4), balance (Biodex SD), and cognitive function (MoCA, Stroop, WAIS-III, TMT), making it one of the few trials to rigorously evaluate physical, cognitive, and dual-task performance outcomes in older adults. This approach is low-cost, scalable, and focused on fall prevention and autonomy maintenance.
  Arms: Pilates

SUMMARY:
Our aims are to evaluate the impact of 24-week combined Pilates and dual-task exercises on physical fitness, balance, cognitive function, bone density in older adults. Participants ≥ 65 years of both genders will be randomly allocated to a control (n= 55) or intervention group (n= 55). Twice a week, sessions will take place in the FADEUP- UPORTO, with moderate intensity Pilates exercise and dual-task exercises. Trunk strength and stability, balance, cognitive function, and physical fitness will be accessed before and after the intervention. The Pilates method is easy to apply, low cost and widely accepted by older adults and it can integrate dual-task exercises easily. The researcher expected the intervention to improve balance, physical and cognitive skills of the participants, which may reduce the number of falls. The investigators seek to contribute with relevant information and enlighten the Dual Task-Pilates program as a safe strategy to reduce falls and maintain elderly's autonomy.

DETAILED DESCRIPTION:
To accomplish our aims the following tasks will be conducted:

1. Disclosure, recruitment and participants characterization (3 months). Participants of both genders, ≥ 65 years old, living in the community, with independent mobility, will be recruited through the "Mais Ativos Mais Vividos" project (in FADEUP), senior universities, and healthcare centers.

   This is a longitudinal experimental study. For sample size, an a priori calculation of statistical power (G*Power 3.1, Dusseldorf, Germany) was performed based on an Ancova. The sample size required to detect an effect size of 0.40; α err prob 0.05 and a power of 0.80 is 111 subjects to accommodate a maximum dropout rate of 20%.
2. Participant´ Assessments (2 months) Participants will be submitted to the following measurements at 2 time points, baseline and post-intervention.

   I - Sociodemographic data and clinical characterization, collected by questionnaire; and health status with Short Form Health Survey (SF-36) II - Weight and height will be measured with a SECA 899 scale and SECA 217 stadiometer (Hamburg, Germany); III - Body composition and bone mineral density will be determined by DEXA, Hologic Explorer QDR 4500 (Bedford, MA / USA); IV - Habitual physical activity assessed by Link ActiGraph GT9X accelerometers for 7 consecutive days (confounder); V - Functional evaluation by the senior fitness test (SFT) including lower (chair stand) and upper (arm curl) limb strength, lower (sit reach) and upper (back scratch) limb flexibility, agility and dynamic balance (timed up and go) and cardiorespiratory endurance (walk 6 min); VI- Handgrip strength with the Jamar analog dynamometer; VII- Balance assessment made in Biodex Balance System SD platform (Biodex Medical Systems, Shirley, NY), including Sensory Integration (CTSIB) and Falls Risk; VIII- Trunk strength assessed using the Biodex System 4 Pro isokinetic dynamometer (Medical Systems, Shirley, NY, USA); IX- Stability of the trunk muscles with Stabilizer Pressure Biofeedback; X- Assessment of cognitive function using the Montreal Cognitive Assessment (MoCA), Trail Making Test (TMT), Stroop Color and Word Test (SCWT), Wechsler Adult Intelligence Scale (WAIS III) e Wechsler Memory Scale (WMS), conducted by an experienced psychologist; XI-Assessment of the cost of dual tasking using the Cognitive timed up ang go.
3. Intervention (5 months) Participants will be allocated to the Experimental Group (EG) and Control Group (CG) in a 1:1 ratio. In the EG, participants will be divided into small groups of 15 to 18 individuals.

   The exercise program, conducted at FADEUP, will run for 20 weeks, consisting of two 60-minute sessions per week at moderate to vigorous intensity. Heart rate monitors (GARMIN Vivosmart 4) and the Borg Rating of Perceived Exertion Scale (1 to 10) will be used to monitor intensity. The program will begin with a 3-week period at light intensity (57% to 63% of maximum heart rate), followed by a progression to moderate intensity (64% to 76%) from weeks 4 to 10, and to moderate-to-vigorous intensity (77% to 95%) from week 11 onward, with increasing complexity of exercises.

   The methodology is based on international training approaches from Polestar® and PhysicalMind® schools. The program includes Pilates exercises designed to improve trunk strength and stability (core), spinal mobility, upper and lower limb strength and flexibility, coordination, balance, agility, control, and concentration. The method emphasizes slow and controlled movements, focusing on both concentric and eccentric phases, with correct posture and movement quality. Dual-task exercises will be integrated into the Pilates routine, combining cognitive activities with physical tasks to promote attention and concentration.

   The selected Pilates exercises include: Cat, Swan, Mermaid, Spine Twist, Spine Stretch Forward, Squat, One Leg Circle, The Roll Down, The Roll Up, The Hundred, Single Leg Stretch, Double Leg Stretch, Bridge, Side Kick, Scissors, Bicycle, Scapular Support, Leg Pull Front, Leg Extension, Swimming, One Leg Kick, and Double Leg Kick. These exercises will be adapted for older adults using chairs, elastic bands, foam rollers, sticks, and balls to increase intensity and complexity.
4. Data analysis and processing Data will be entered into a database using SPSS (Statistical Package for the Social Sciences, version 29) and subsequently processed and analyzed. Descriptive statistics will be presented as medians and interquartile ranges or means and standard deviations, as well as counts and percentages, as appropriate. ANCOVA and repeated measures ANOVA will be used to compare differences between groups and time points. A 95% confidence interval will be applied. Only data from participants with an attendance rate of 75% or higher will be included in the analysis.
5. Dissemination of results This intervention is part of a doctoral project and will adhere to the principles of the Declaration of Helsink and the National Legislation. The results will be disseminated through four scientific articles and presentations at national and international conferences related to the study themes: physical and cognitive activity in older adults, Pilates, and fall risk.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (≥ 60 years)
* Both sexes
* Healthy (no diseases or diagnoses that prevent physical exercise)
* Community-dwelling

Exclusion Criteria:

* Individuals diagnosed with medical conditions for which physical activity is not recommended, including, but not limited to, musculoskeletal problems, cardiovascular diseases, and/or severe respiratory diseases.
* Participants with neurological diseases or disabling conditions that compromise balance.
* Individuals with moderate or severe cognitive impairment, according to established normative test values.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Balance- Biodex balance System SD | Baseline, post 20 weeks.
  The Biodex Balance System SD plataform was used to assess balance through the Sensory Integration Test (CTSIB) and the Falls Risk Test. These assessments evaluate how the central nervous system processes sensory inputs (visual, and proprioceptive systems) to maintain postural control, helping to identify balance impairments and fall risk (Biodex Medical Systems, Shirley, NY).
Stability of the trunk muscles- Stabilzer Pressure Biofeedback Unit | Baseline, post 20 weeks
  The study by Grooms et al. (2013) evaluated trunk muscle stability using the Stabilizer Pressure Biofeedback Unit, a device that measures the activation of deep abdominal muscles during exercises. It helps ensure proper engagement of core stabilizers, such as the transversus abdominis and multifidus, making it useful for both assessment and rehabilitation.
Balance- Single-Leg Stance Test | Baseline, post 20 weeks.
  The Single-Leg Stance Test is a simple and widely used method for assessing static postural balance. It involves standing on one leg, with eyes open, for up to 45 seconds. This test has been validated by Springer et al. (2007), who demonstrated its reliability in detecting balance deficits and fall risk, particularly in older adults and clinical populations.
Functional Fitness (Strength)- SFT | Baseline, 20 weeks.
  The Senior Fitness Test includes specific assessments for upper and lower body strength in older adults. Lower body strength is measured using the 30-second chair stand test, which evaluates leg strength and endurance. Upper body strength is assessed with the 30-second arm curl test, measuring arm muscle strength. These tests were validated by Rikli and Jones (1999) and are considered reliable indicators of functional fitness in elderly populations.
Functional Fitness (Flexibility)- SFT | Beseline, post 20 weeks.
  The Senior Fitness Test includes two flexibility assessments aimed at older adults: the Sit and Reach Test, which evaluates lower body flexibility, particularly of the hamstrings and lower back; and the Back Scratch Test, which assesses upper body flexibility, focusing on shoulder mobility. Both tests were validated by Rikli and Jones (1999) and are widely used to detect limitations in functional range of motion.
Cardiorespiratory endurance- SFT | Baseline, post 20 weeks.
  The 6-Minute Walk Test is part of the Senior Fitness Test and evaluates cardiorespiratory endurance in older adults. Participants are instructed to walk as far as possible in six minutes along a 50-meter rectangular course. This test was validated by Rikli and Jones (1999) and is considered an excellent indicator of functional capacity for daily activities, such as climbing stairs or performing household tasks.
Dynamic balance and agility- 8-Foot Up-and-Go Test | Baseline, post 20 weeks.
  The 8-Foot Up-and-Go Test is part of the Senior Fitness Test and assesses agility and dynamic balance in older adults. The participant must stand up from a chair, walk 2.44 meters (8 feet) quickly, turn around a cone, and return to the seat as fast as possible (Rikli and Jones, 1999).
Handgrip strength | Baseline, 20 weeks.
  Handgrip strength was assessed using the Jamar analog dynamometer (Sammons Preston Inc., Bolingbrook, Illinois, USA), a gold-standard instrument widely used to measure upper limb strength. The test is simple, quick, and provides a reliable indicator of overall functional strength. The Jamar dynamometer has well-established validity in clinical research.
Trunk strength- Biodex System 4 Pro isokinetic dynamometer | Baseline, 20 weeks
  Trunk strength was assessed using the Biodex System 4 Pro isokinetic dynamometer (Biodex Medical Systems, Shirley, NY, USA), a highly accurate device used to measure muscular torque and power at various speeds. It is widely used in clinical and research settings to analyze muscular performance in a standardized and safe manner.

SECONDARY OUTCOMES:
Cognitive function- MoCA | Baseline, 20 weeks.
  Cognitive function was assessed using the Montreal Cognitive Assessment (MoCA), a brief and validated tool for screening mild cognitive impairment. The test evaluates multiple cognitive domains, including memory, attention, language, visuospatial abilities, and executive function. The MoCA is sensitive for detecting early cognitive decline in older adults (Nasreddine, Z. S., et al., 2005).
Cognitive function- Trail Making Test | Baseline, 20 weeks.
  Executive cognitive function was assessed using the Trail Making Test (TMT), parts A and B. Part A evaluates visual attention and processing speed, while part B measures cognitive flexibility and executive control, requiring alternating between numbers and letters. The TMT is widely used and validated for detecting cognitive impairment in older adults (Reitan, R. M., 1958).
Cognitive function- Stroop Color and Word Test | Baseline, 20 weeks.
  The Stroop Color and Word Test (SCWT) was employed to assess cognitive inhibition and selective attention. The test includes reading color words, naming ink colors, and naming ink colors when the word and ink are incongruent. This version follows Bickford et al. (2018) and is sensitive to detecting cognitive interference, making it valuable in clinical settings to identify executive dysfunction.
General intelligence- Wechsler Adult Intelligence Scale (WAIS-III) | Baseline, 20 weeks
  General intelligence was assessed using the WAIS-III, a standardized scale that measures various cognitive domains in adults, including verbal comprehension, perceptual reasoning, working memory, and processing speed. It is widely recognized for its validity and reliability in the assessment of intellectual functioning (Wechsler, D., 1997).
Cognitive function- Memory function | Baseline, 20 weeks.
  Memory function was assessed using the Wechsler Memory Scale (WMS), a validated tool that evaluates immediate and delayed memory, attention, and learning ability. It is commonly used in clinical settings to diagnose memory disorders and monitor cognitive changes over time (Wechsler, D., 1997).
Sociodemographic questionnaire and and clinical characterization | Baseline, 20 weeks.
  Sociodemographic questionnaire which includes the following variables: ID, group allocation, birth date, age, sex, education level, profession, number of falls, diagnosed diseases. Quality of life satisfaction will also be evaluated using self-report.
Height assessment | Baseline, 20 weeks
  Height was measured using the Seca 217 mobile stadiometer, with participants standing upright and barefoot. Measurements were recorded in centimeters.
Body mass | Baseline, 20 weeks.
  Body mass (kg), fat-free mass (kg), fat mass (kg) and BMI will be analyzed with bioimpedance (InBody 120®).
Bone mineral density | Baseline, 20 sections
  Bone mineral density will be assessed by DEXA (Hologic QDR Explorer 4500, Bedford, MA, USA) at the lumbar spine and femoral neck.

OTHER OUTCOMES:
Habitual physical activityBaseline, 20 weeks. | Baseline, 20 weeks.
  Habitual physical activity will be assessed using ActiGraph GT9X Link accelerometers worn for 7 consecutive days.

CONTACTS AND LOCATIONS:
Overall Officials: Joana Carvalho, PhD, Study Director — CIAFEL
Locations (1):
- CIAFEL, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No
Data management will comply with applicable data protection legislation and the internal guidelines of the University of Porto. All project-specific documents, including collected data, will be stored with full privacy and confidentiality, with access restricted to the principal investigator and their advisors. The data will be destroyed after the objectives of the study are fulfilled or after five years, whichever comes first. All information obtained through questionnaires and direct observation will be anonymized before storage.

REFERENCES:
- [Background] García-Vaquero, M. P., García-Manso, J. M., Pérez-López, J., Olcina, G., & Molinero, O. (2016). Reliability and learning effects of an isokinetic trunk extension-flexion protocol using the Biodex System 4. Clinical Biomechanics, 31, 627-630. https://doi.org/10.1016/j.clinbiomech.2016.05.003
- [Background] Reitan, R. M. (1958). Validity of the Trail Making Test as an Indicator of Organic Brain Damage. Perceptual and Motor Skills, 8(3), 271-276. https://doi.org/10.2466/pms.1958.8.3.271 (Original work published 1958)
- [Background] Stroop, J. R. (1935). Studies of interference in serial verbal reactions. Journal of Experimental Psychology, 18(6), 643-662. https://doi.org/10.1037/h0054651
- [Background] Intertester and intratester reliability of a dynamic balance protocol using the Biodex Stability System. Journal of Sport Rehabilitation, 7(2), 95-101. https://doi.org/10.1123/jsr.7.2.95
- [Background] Springer BA, Marin R, Cyhan T, Roberts H, Gill NW. Normative values for the unipedal stance test with eyes open and closed. J Geriatr Phys Ther. 2007;30(1):8-15. doi: 10.1519/00139143-200704000-00003. PMID 19839175
- [Background] Wechsler, D. (1997). WAIS-III: Wechsler Adult Intelligence Scale - Third Edition Manual. San Antonio, TX: The Psychological Corporation.
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019